CLINICAL TRIAL: NCT03640637
Title: Accuracy of PET/MRI in Diagnosis and Treatment Evaluation of Children and Adolescents With Inflammatory Bowel Disease
Brief Title: The Role of PET/MRI in the Diagnosis and Treatment of Children and Adolescents With Inflammatory Bowel Diseases
Acronym: PEDICAD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Steffen Husby, Professor, MD, DMSc, Odense University Hospital
Other Study IDs: OUH-HCA-003
Record Dates: First submitted 2018-08-15; First posted 2018-08-21 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Positron emission tomography; Magnetic resonance imaging
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suspected IBD: A prospective study of 50 pediatric patients suspected of IBD. Participants will undergo routine diagnostic procedures for evaluation of pediatric IBD including blood samples, faecal samples, endoscopies (colonoscopy and gastroscopy with biopsy/histology) and MRI of the abdomen. In addition, a PET scan will be performed in this protocol and combined with MRI. For accuracy measures, PET/MRI scan will be compared to the combined findings of endoscopy, histology and severity of inflammation by clinical scoring systems (weighted Pediatric Crohn's Disease Activity Index (wPCDAI) for CD and Pediatric Ulcerative Colitis activity Index (PUCAI) for CU), faecal calprotectin and biochemistry.
- Treatment response group: A pilot study of 10-15 patients previously diagnosed with CD who will undergo PET/MRI scan as an investigational procedure before initiation of biological treatment with an anti-TNF-alpha antibody (infliximab, adalimumab) because of disease relapse or steroid dependent disease. Patients will be scheduled for a PET/MRI again after one month. This study will evaluate if PET/MRI can diagnose a flare in CD and if PET/MRI is a reliable imaging tool to monitor intestinal inflammation. In this study the patient will act as his/her own control.

SUMMARY:
The purpose of this study is to test the utility of PET/MRI in diagnosis and management of Inflammatory bowel disease (IBD) in children and adolescents, hereby

* To test if PET/MRI scan is an accurate method to diagnose and differentiate Crohn's disease and Ulcerous Colitis in children and adolescents suspected of IBD.
* To evaluate whether PET/MRI scan in children and adolescents with Crohn's disease is an accurate method to diagnose relapses and to monitor the effect of biological treatment with monoclonal antibodies directed towards Tumor Necrosis Factor-alpha.

DETAILED DESCRIPTION:
Crohn's disease and Ulcerous Colitis constitute the primary inflammatory bowel diseases. Crohn's disease can affect any part of the digestive tract, from mouth to anus, and inflammation can be present in all layers of the intestinal wall. Ulcerous Colitis is primarily located in the inner layer of the colonic bowel wall.

In the pediatric population, current diagnostic strategies involve blood tests, fecal sampling (calprotectin), magnetic resonans (MRI) scan and both upper and lower endoscopies. In this population endoscopy requires general anesthesia and involves the risk of bowel wall perforation.

A known method of identifying inflammation is by Positron Emission Tomography (PET). In this procedure a radioactively labelled sugar molecule is injected into the blood stream via a venous catheter. The inflammatory cells take op relatively more of the sugar, compared to normal cells, and the cells are visible on the scan. Until now the anatomic localization of the inflammation has been poor but recently is has become possible to combine the MRI scan with PET resulting in excellent localization, with minimal radiation exposure (corresponding to 1 year background radiation in Denmark).

To make diagnosis and identification of inflammation flares during treatment safer for children and adolescents we aim to investigate whether PET/MRI is accurate in diagnosing IBD in children and adolescents and in diagnosing flares in children with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Suspected of having IBD
* Planned to undergo standard evaluation OR
* Known Crohn's disease about to start anti-TNF therapy due to steroid dependency or disease relapse.

Exclusion Criteria:

* Active or prior diagnosis of inflammatory disease other than IBD
* Active or prior diagnosis of cancer
* Type 1 diabetes
* Not able to lie still for the MRI scan.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (aged 8-17) referred from general practice to pediatric evaluation for IBD at tertiary centres, either H. C. Andersens Childrens Hospital, Odense University Hospital or Department of Pediatrics, Lillebaelt Hospital OR children with known Crohn's disease about to start anti-TNF therapy.
  Adolescents (aged 18-25) referred from general practice to evaluation for IBD at the Department of Gastroenterology, Odense University Hospital OR adolescents about to start anti-TNF therapy.
  Newly diagnosed patient, who start anti-TNF therapy at inclusion will be included in both studies.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, accuracy and predictive value of PET/MRI at diagnosis of IBD and in differentiating Crohn's disease and Ulcerous colitis. | 6 months
  PET/MRI will be compared to standard evaluation: Clinical symptom scoring systems (for Crohns disease: wPCDAI, for Ulcerous colitis: PUCAI), faecal calprotectin, C-reactive protein and endoscopy with histology.
  Endoscopy will be used for gold reference. PET/MRI scans will be analysed for PET uptake values pr. bowel segment for each patient and compared to standard evaluation results.
Sensitivity, specificity and accuracy of PET/MRI in diagnosing disease flare in Crohn's disease and to evaluate inflammatory response to anti-TNF treatment. | 1 month
  PET/MRI will be compared to standard evaluation: Clinical symptom scoring systems (wPCDAI), faecal calprotectin, C-reactive protein and endoscopy with histology.
  The patient will serve as his/her own control. This will be a pilot study. PET/MRI scans will be analysed for PET uptake values pr. bowel segment for each patient and compared to standard evaluation results.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Husby, Professor, Principal Investigator — Odense University Hospital
Locations (1):
- Steffen Husby, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Project data management plan is still being developed.